CLINICAL TRIAL: NCT02508883
Title: Comparison Among the Scores of Glasgow-Blacthford, Rockall and AIMS65 for the Prediction of Rebleeding and Mortality in Patients With Cancer and Upper Gastrointestinal Bleeding
Brief Title: Evaluation of Prognostic Scores in Patients With Upper Gastrointestinal Bleeding and Cancer
Status: Completed | Type: Observational
Sponsor: Instituto do Cancer do Estado de São Paulo (Other)
Responsible Party: Sponsor
Other Study IDs: NP621/14
Record Dates: First submitted 2015-05-29; First posted 2015-07-27 (Estimated); Last update posted 2016-10-06 (Estimated); Status verified 2016-10

CONDITIONS: Upper Gastrointestinal Bleeding
Keywords: Cancer; hemorrhage; endoscopy; gastrointestinal hemorrhage
MeSH Terms: conditions — Gastrointestinal Hemorrhage; Neoplasms; Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Upper gastrointestinal bleeding: patients with cancer who presented or were admitted in the emergency room, wards or intensive care units of the Cancer Institute of São Paulo (ICESP), with a recent episode of upper gastrointestinal bleeding.

SUMMARY:
This is a prospective and observational study to evaluate oncologic patients that presented upper gastrointestinal bleeding with the use of some prognostic scores.

DETAILED DESCRIPTION:
Background: Cancer incidence is rising worldwide, therefore complications of this condition, such as bleeding, are also expected to be more frequently seen.

Tumoral bleeding is usually difficult to control and the bleeding episode may represent the end stage of the malignant disease. In this context, it is relevant to study the performance of prognostic scores to prediction of clinical outcomes in patients with cancer.

Objective: To evaluate and compare the performance of prognostic scores to predict clinical outcomes in a group of patients with cancer of any site that has presented a recent episode of upper gastrointestinal bleeding (UGIB).

Design: Prospective and observational study. Setting: Cancer Institute of São Paulo; University of são Paulo. Patients: All patients with cancer referred to the Endoscopy Unit because of upper gastrointestinal bleeding will be included consecutively.

Main Outcome Measurements: need and amount of blood transfusions administered, need for endoscopic therapy, surgery, rebleeding, and mortality at 30 days.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of malignant neoplasm of any site, either located inside or outside of GI tract;
* Current evidence of bleeding in the last 48 hours, either by presenting hematemesis and/or melena, with or without hemodynamic instability. Patients with hematochezia or bright red blood per rectum due to a site of bleeding in upper GI tract will also be included.

Exclusion Criteria:

* Age < 18 years-old;
* Suspicion or confirmation of pregnancy.
* Patients with no evidence of malignant neoplasm after curative surgery or oncologic therapy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients referred to the Endoscopy Unit of ICESP because of upper gastrointestinal bleeding will be included consecutively, according to the selection criteria mentioned below.
  The analysis of our recent data base allows us to estimate an accrual of about 300 patients at the end of 1 year of study.
Sampling Method: Probability Sample
Enrollment: 243 (Actual)
Dates: Start 2015-04; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
blood transfusions administered | 30 days
  The need and amount of blood transfusions administered
Endoscopic therapy | 30 days
  Hemostatic endoscopic therapy will be performed if there are findings of active or recent bleeding, under conscious or deep sedation after hemodynamic stabilization and oral fasting
Surgery | participants will be followed for the duration of hospital stay, an expected average of 30 days
  need for surgery to control tumour bleeding
rebleeding | 30 days
  episodes of rebleeding
mortality | 30 days
  mortality

SECONDARY OUTCOMES:
Finding the cut-off value of highest sensitivity and specificity of Rockall, Glasgow-Blatchford and AIMS65 scores employing the receiver operating curve (ROC). | 1 year
  find the cut-off value of highest sensitivity and specificity of Rockall, Glasgow-Blatchford and AIMS65 scores for discriminant selection of a low-risk group, if one exists, among patients with recent upper gastrointestinal bleeding and cancer with confirmed diagnosis, located inside or outside the GI tract, who could be managed on an outpatient basis.

CONTACTS AND LOCATIONS:
Overall Officials: Fauze Maluf-Filho, MD, PHD, Principal Investigator — Cancer Institute of São Paulo
Locations (1):
- Cancer Institute of São Paulo, São Paulo, São Paulo, Brazil